CLINICAL TRIAL: NCT04182841
Title: RheOx European Post-Market Clinical Study
Brief Title: RheOx Registry Study in Europe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gala Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS005
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Chronic Bronchitis; COPD
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: RheOx Treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- RheOx Treatment (Other): RheOx is a CE-marked device-based, energy delivery system that delivers energy to ablate soft tissue such as the airway epithelium and sub-mucosal tissue layers. The energy is delivered via a proprietary catheter through the bronchoscope.
  Interventions: Device: RheOx

INTERVENTIONS:
Device: RheOx — RheOX is a CE-marked device-based, energy delivery system that delivers energy to ablate soft tissue such as the airway epithelium and sub-mucosal tissue layers. The energy is delivered via a proprietary catheter through the bronchoscope.

SUMMARY:
Post-market clinical study (registry study) to collect post-market safety and clinical utility data in European patients with chronic bronchitis treated with RheOx.

DETAILED DESCRIPTION:
RheOx is a device-based, energy delivery system that delivers high frequency short duration energy to the airway epithelium and sub-mucosal tissue layers. The energy is delivered via a proprietary catheter through the bronchoscope.

Two sessions of treatment will be delivered one month apart. The right lung is treated at the first treatment session and the left lung is treated at the second treatment session (approximately one month after the right side is treated). Treatment will be delivered by a respiratory physician (interventional pulmonologist) in a tertiary teaching hospital during a bronchoscopic procedure. The bronchoscopy will be delivered during general anaesthesia. It is anticipated that the bronchoscopic procedure will last less than 60 minutes in total. Treatment will be deemed to have been delivered following the successful treatment during the two bronchoscopies.

Subjects will be required to submit to several tests and questionnaires during the study including respiratory function tests.

ELIGIBILITY:
Inclusion Criteria:

* Patient has moderate to severe Chronic Bronchitis

Exclusion Criteria:

* Patient has an implantable cardioverter defibrillator, pacemaker, or any other implantable electronic device.
* Patient has history of ventricular tachyarrhythmia or any clinically significant atrial tachyarrhythmia (i.e., abnormality with vital signs) and/or history of type II second or third degree AV block.
* Patient has airway stent(s), valves, coils, or other lung implant/prosthesis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of SAEs | Through end of study (24 months post bilateral treatment)
  Incidence of serious adverse events associated with RheOx treatment through 24 months
Quality of Life: CAT | Through end of study (24 months post bilateral treatment)
  COPD Assessment Test (CAT) questionnaire
Quality of Life: SGRQ | Through end of study (24 months post-bilateral treatment)
  St. George Respiratory Questionnaire

SECONDARY OUTCOMES:
Pulmonary Function: FEV1 | Through end of study (24 months post-bilateral treatment)
  Forced expiratory volume (FEV). FEV1 is the amount of air you can force from your lungs in one second.
Pulmonary Function: FVC | Through end of study (24 months post-bilateral treatment)
  Forced Vital Capacity
COPD Exacerbations | Through end of study (24 months post-bilateral treatment)
  COPD Exacerbations

CONTACTS AND LOCATIONS:
Overall Officials: William Krimsky, MD, Study Director — Gala Therapeutics, Inc.
Locations (2):
- Otto Wagner Spital, Vienna, Austria
- Pneumologie Thoraxklinik Heidelberg gGmbH University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No